CLINICAL TRIAL: NCT00315809
Title: Molecular Epidemiology of Leprosy - Philippines
Status: Completed | Type: Observational
Sponsor: Colorado State University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Varalakshmi Vissa, Colorado State University
Other Study IDs: 05-0080
Record Dates: First submitted 2006-04-17; First posted 2006-04-19 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: Leprosy
Keywords: leprosy, Philippines
MeSH Terms: conditions — Leprosy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to see if new methods can be used to determine why Multidrug Therapy (MDT), used to cure leprosy patients effectively for twenty years, is not as effective against Leprosy in the Philippines. Researchers do not know how people get infected with leprosy or what causes the disease to relapse after cure with adequate MDT. Blood, skin scrapings, nasal swabs and biopsies, will be collected from leprosy patients to perform tests related to the detection of the disease and the germ. The tests will be used to find out if the bacteria in the body are related to the bacteria found in other patients or contacts. This will help the researchers to know where these bacteria come from, and to see how they spread. Other tests will be performed to see if the bacteria can be killed by two common medicines given to leprosy patients. Study participants will include individuals age 18 and older presenting to Leonard Wood Memorial for the diagnosis and/or relapse of leprosy.

DETAILED DESCRIPTION:
The overall objectives of this study are to understand the factors leading to continued incidence of leprosy in the Philippines by novel molecular methodologies using a combination of retrospective and prospective sampling approaches. The overall objectives include: (1) strain typing of M. leprae isolates obtained from new and relapsed leprosy patients in the Philippines to identify clusters and transmission patterns when combined with conventional epidemiological criteria; (2) to determine the viability of M. leprae by mRNA detection in specimens collected from new patients; and those with signs of relapse; (3) to identify and determine the extent of mutations conferring resistance in past and circulating M. leprae isolates from leprosy patients to two Multidrug therapy (MDT) drugs; Dapsone and Rifampicin and; (4) to detect chains of transmission in endemic populations by a retrospective analyses of isolates in sample banks when combined with strain typing information from new cases and conventional epidemiological criteria. The following are the outcome measures for each of the objectives: (1) strain typing: identification of genotypes; (2) percent of samples from patients and their contacts containing viable M. leprae (as judged by the presence of mRNA for a panel of M. leprae genes; (3) percent of samples from patients and their contacts containing mutations in M. leprae rpoB and folP 1 genes and identification of new mutations associated with relapse and; (4) identification of matching or similar genotypes in new samples obtained from patients and their household contacts with those in retrospective samples. Clinical specimens that contain M. leprae bacilli such as skin biopsy, slit skin smears, nasal swabs and blood are required to obtain M. leprae DNA to meet the objectives of the study. Nasal swabs will be used for assessing the role of the nasal mucosa in infection and dissemination in leprosy. The blood is useful for monitoring the humoral responses to infection. Skin biopsy, slit skin smears, nasal swabs and blood will be obtained from informed consenting patients. Enrollment and sample collection procedures will take approximately 1-2 hours. These procedures will be performed during the patient's visit to the clinic for diagnosis and therapy for leprosy. As part of the study, a punch biopsy from a lesion is being collected to enable sufficient quantities of DNA to be extracted for strain typing, a critical objective of this study. Patients will be required to visit the site once more after 7-10 days to assess the biopsy site. This visit may take 30-60 minutes. An epidemiology survey containing demographic and clinical information will be obtained from each participant. Study participants for prospective sample collections will include volunteering and consenting individuals, 18 years old and above, reporting at Leonard Wood Memorial (LWM) CebuSkin Clinic, Leonard Wood Memorial Center for Biomedical Research, Cebu, Philippines for the diagnosis of leprosy and/or relapse of leprosy.

ELIGIBILITY:
Inclusion Criteria:

1. All Leprosy patients eighteen years and above who are consulting at the LWM will be invited to participate.

Exclusion Criteria:

1. Patients unwilling to participate or unable to give informed consent will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Blood, nasal swabs, slit skin smears and biopsies will be obtained prospectively from individuals greater than 18 years of age, representing newly diagnosed and relapse leprosy patients. The study participants will be obtained from LWM clinic. DNA and RNA based methodologies will be developed and applied to obtain data necessary for substantiation of a number of factors implicated in transmission of leprosy in Philippines.
Sampling Method: Non-Probability Sample
Enrollment: 310 (Actual)
Dates: Start 2006-04; Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Varalakshmi D Vissa, PhD, Study Director — Colorado State University; Maria Felicio-Balagon, MD, Principal Investigator — Leonard Wood Memorial, Cebu, Phillippines
Locations (1):
- Leonard Wood Memorial Center, Cebu City, Philippines

REFERENCES:
- [Background] Kimura M, Sakamuri RM, Groathouse NA, Rivoire BL, Gingrich D, Krueger-Koplin S, Cho SN, Brennan PJ, Vissa V. Rapid variable-number tandem-repeat genotyping for Mycobacterium leprae clinical specimens. J Clin Microbiol. 2009 Jun;47(6):1757-66. doi: 10.1128/JCM.02019-08. Epub 2009 Apr 22. PMID 19386839
- [Result] Sakamuri RM, Kimura M, Li W, Kim HC, Lee H, Kiran MD, Black WC 4th, Balagon M, Gelber R, Cho SN, Brennan PJ, Vissa V. Population-based molecular epidemiology of leprosy in Cebu, Philippines. J Clin Microbiol. 2009 Sep;47(9):2844-54. doi: 10.1128/JCM.02021-08. Epub 2009 Jul 1. PMID 19571027